CLINICAL TRIAL: NCT01845896
Title: Rehabilitation in MS: Influence of High Intensity Exercise on Insulin Resistance, Muscle Contractile Properties, Aerobic Capacity and Body Composition in Multiple Sclerosis
Brief Title: Influence of High Intensity Exercise on Insulin Resistance, Muscle Contractile Properties, Aerobic Capacity and Body Composition in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bert Op't Eijnde (Other)
Responsible Party: Sponsor-Investigator, Bert Op't Eijnde, Ph.D, Hasselt University
Organization: Hasselt University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13.20/reva13.02
Record Dates: First submitted 2013-04-30; First posted 2013-05-03 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Multiple Sclerosis; Healthy Controls
Keywords: high intensity interval training; combined training; insulin resistance; muscle contractile properties
MeSH Terms: conditions — Multiple Sclerosis; Insulin Resistance | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Combined exercise (Experimental): 12 weeks combined exercise programme (supervised)
  Interventions: Behavioral: Training
- High intensity interval training (Experimental): 12 weeks high intensity interval exercise programme (supervised)
  Interventions: Behavioral: Training
- Control (No Intervention): sedentary/habitual lifestyle

INTERVENTIONS:
Behavioral: Training
  Other Names: 12 weeks of high intensity interval training or combined exercise
  Arms: Combined exercise; High intensity interval training

SUMMARY:
The purpose of this study is to investigate the effects of a combined training programme and a high intensity interval training programme on insulin resistance, muscle strength/ muscle contractile properties, aerobic capacity and body composition in MS patients.

It is assumed that the the above mentioned clinical parameters will improve due to physical exercise.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed MS according to the McDonald criteria
* Expanded Disability Status Scale (EDSS) between 0.5 and 6
* Be able to train 5 times in 2 weeks at the University

Exclusion Criteria:

* Comorbidities like cardiovascular-, respiratory-, orthopaedic or metabolic diseases (like diabetes type 2)
* Having had an relapse in a period of 3 months prior to the start of the intervention period
* Having an relapse during the intervention period
* Pregnancy and other contra indications for physical activity
* Mental disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
insulin sensitivity (insulin profile) | change from baseline to 12 weeks
  glucose and insulin concentration measurements in blood
muscle contractile properties | from baseline to 12 weeks
  measurements of cross sectional area and fiber distribution in muscle fibers of the m. vastus lateralis + measurements of enzymatic reactions, ATP, glycogen, ...

SECONDARY OUTCOMES:
muscle strength of knee extensor/flexor | change from baseline to 12 weeks
  by means of an isokinetic dynamometer the muscle strength and endurance will be measured
aerobic capacity | change from baseline to 12 weeks
  by means of a submaximal endurance test (ergometer)
cytokine profile | change from baseline to 12 weeks
  measurements of blood cytokine levels
Self-reported measures | Change from baseline to 12 weeks
  The self-reported measures contains some questionnaires
body composition | Change from baseline to 12 weeks
  Weight, body fat% and lean tissue% will be assessed by means of a DEXA scan

CONTACTS AND LOCATIONS:
Overall Officials: Inez Wens, M.Sc., Principal Investigator — Reval/Biomed, Hasselt University; Bert Opt Eijnde, Ph.D, Study Chair — Reval/Biomed, Hasselt University
Locations (1):
- Reval, Diepenbeek, Belgium

REFERENCES:
- [Derived] Wens I, Dalgas U, Vandenabeele F, Grevendonk L, Verboven K, Hansen D, Eijnde BO. High Intensity Exercise in Multiple Sclerosis: Effects on Muscle Contractile Characteristics and Exercise Capacity, a Randomised Controlled Trial. PLoS One. 2015 Sep 29;10(9):e0133697. doi: 10.1371/journal.pone.0133697. eCollection 2015. PMID 26418222
- [Derived] Hansen D, Wens I, Vandenabeele F, Verboven K, Eijnde BO. Altered signaling for mitochondrial and myofibrillar biogenesis in skeletal muscles of patients with multiple sclerosis. Transl Res. 2015 Jul;166(1):70-9. doi: 10.1016/j.trsl.2015.01.006. Epub 2015 Jan 20. PMID 25666356
- [Derived] Wens I, Dalgas U, Vandenabeele F, Krekels M, Grevendonk L, Eijnde BO. Multiple sclerosis affects skeletal muscle characteristics. PLoS One. 2014 Sep 29;9(9):e108158. doi: 10.1371/journal.pone.0108158. eCollection 2014. PMID 25264868